CLINICAL TRIAL: NCT02433626
Title: A Phase 1 Study of COTI-2 as Monotherapy or Combination Therapy for the Treatment of Advanced or Recurrent Malignancies
Brief Title: Study of COTI-2 as Monotherapy or Combination Therapy for the Treatment of Malignancies
Acronym: COTI2-101
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Critical Outcome Technologies Inc. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other); Northwestern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COTI2-101
Record Dates: First submitted 2015-04-27; First posted 2015-05-05 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Endometrial Cancer; Cervical Cancer; Peritoneal Cancer; Head and Neck Cancer; HNSCC; Colorectal Cancer; Lung Cancer; Pancreatic Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Lung Neoplasms; Pancreatic Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COTI2 (Experimental): COTI-2 will be self-administered as a single agent, orally, once daily for 5 days followed by 2 treatment-free days each week; 1 cycle will be defined as 4 weeks of treatment as described (5 days on, 2 days off per week). Participants will remain on treatment until they experience a lack of benefit.
  Interventions: Drug: COTI2
- COTI2 + cisplatin (Experimental): COTI-2 will be self-administered as a single agent, orally, once daily for 5 days followed by 2 treatment-free days each week; 1 cycle will be defined as 3 weeks of treatment as described (5 days on, 2 days off per week). Cisplatin 60 mg/m2 IV will be administered on Day 1 of each 3 week cycle. Participants will remain on treatment until they experience a lack of benefit.
  Interventions: Drug: COTI2; Drug: Cisplatin

INTERVENTIONS:
Drug: COTI2 — COTI-2 is a third generation thiosemicarbazone.
  Other Names: CAS 1039455-84-9; 4-(2-pyridinyl)-2-(6,7-dihydro-8(5H)-quinolinylidene)hydrazide-1-piperazinecarbothioic acid
Drug: Cisplatin — Cisplatin is approved to treat a range of solid tumors and lymphomas.
  Other Names: CAS 15663-27-1; CDDP
  Arms: COTI2 + cisplatin

SUMMARY:
Activity of COTI-2 has been demonstrated in various cancer tumor models. With its p53- and AKT-based mechanisms of action, COTI-2 is anticipated to be highly relevant in treatment of patients with gynecologic malignancies or head and neck squamous cell carcinoma (HNSCC) as well as a variety of other tumor types.

This study is designed primarily to assess the safety and tolerability of COTI-2 monotherapy or combination therapy in patients with advanced and recurrent malignancies to establish a recommended Phase 2 dose (RP2D) for future studies.

Patients are currently being recruited for Part 3 of the study.

Critical Outcome Technologies Inc. has been renamed to Cotinga Pharmaceuticals.

DETAILED DESCRIPTION:
This is a three-part, multi-center, open-label, Phase 1, first-in-patient study of COTI-2 in patients with recurrent ovarian, fallopian tube, primary peritoneal, endometrial, or cervical cancer (collectively gynecological malignancies), and in patients with head and neck squamous cell carcinoma (HNSCC), colorectal, lung, or pancreatic cancer. Other tumor types may be allowed with Sponsor approval.

COTI-2 will be self-administered as a single agent, orally, once daily for 5 days followed by 2 treatment-free days each week.

Part 1 of the study will be dose finding in patients with gynecological malignancies using a 3 + 3 design to establish the MTD (maximum tolerated dose) over 6 planned cohorts.

Part 2 of the study will be dose finding in patients with HNSCC using a 3 + 3 design to establish the MTD over 6 planned cohorts.

Part 3 of the study will be dose finding for COTI-2 in combination with cisplatin in patients with gynecological malignancies, HNSCC, colorectal, lung, pancreatic cancer, or other tumor types with Sponsor approval.

ELIGIBILITY:
Inclusion Criteria

1. ≥18 years of age.
2. Willing and able to provide written informed consent to participate in this investigational study.
3. Cancer that is recurrent, metastatic, or unresectable and for which no effective or curative measures exist.

   * Part 1: Ovarian, fallopian tube, primary peritoneal, endometrial, or cervical cancer
   * Part 2: HNSCC, with confirmed p53 mutations
   * Part 3: Gynecological malignancies, HNSCC, colorectal, lung, pancreatic cancer, or other tumors with Sponsor approval.
4. Ability to attend all scheduled study visits
5. Measurable disease by physical examination or imaging as defined by RECIST v1.1 criteria or evaluable disease as defined by Gynecologic Cancer Intergroup (GCIG) CA125 criteria.
6. European Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Life expectancy ≥3 months.
8. Adequate bone marrow, liver, renal, and cardiac function at study entry, assessed as follows:

   * Hemoglobin ≥9.0 g/dL;
   * Absolute neutrophil count (ANC) ≥1.5 x 109/L;
   * Platelet count ≥100 x 109/L;
   * Prothrombin time (PT) or international normalize rate (INR) within 1.5x upper limit of normal;
   * Partial thromboplastin time (PTT) within 1.5x upper limit of normal;
   * Total bilirubin within normal limits;
   * Alanine transaminase (ALT) and aspartate transaminase (AST) within 1.5x upper limit of normal;
   * Calculated creatinine clearance >50 mL/min;
   * Urine protein <500 mg or urine protein: creatinine ratio (UPC) <1.0; and
   * Left ventricular ejection fraction (LVEF) ≥55% (or the institutional lower limit of normal [LLN]) as evidenced on ECHO.
9. Prior chemotherapy, other investigational agents, or radiation must be discontinued for at least 28 days prior to the first administration of COTI-2. Hormone treatments must be discontinued for at least 28 days prior to the first administration of COTI-2.
10. Toxicity from prior therapy (except alopecia) has resolved to ≤Grade 1; in the event of toxicity that has not resolved to ≤Grade 1 but is considered stable, the patient may be eligible after discussion among the investigator and sponsor's medical monitor.
11. Physiologically incapable of becoming pregnant, postmenopausal, or negative pregnancy test and agree to use adequate contraception (e.g., oral contraceptive, double barrier method, intra-uterine device, intra-muscular contraceptive).
12. Patients enrolled in the expansion phase must be willing to undergo pre and post-Cycle 1 biopsies.
13. Patients enrolled in the escalation and expansion phases will be required to have archival tissue available for analysis.

Exclusion Criteria:

1. Pregnant or lactating.
2. History of other invasive malignancies, with the exception of non-melanoma skin cancer or successfully treated in situ carcinoma, if there is evidence of the malignancy being present within the last 3 years.
3. Inability to tolerate oral medications.
4. Any serious and/or unstable pre-existing medical, psychiatric, or other condition (e.g., severe hepatic impairment) or current unstable or uncompensated respiratory or cardiac conditions which makes it undesirable for the patient to participate in the study or which could jeopardize compliance with the protocol.
5. History of clinically significant or uncontrolled cardiac disease including but not limited to:

   1. Myocardial infarction,
   2. Angina pectoris,
   3. Congestive heart failure of New York Heart Association (NYHA) Grade >2,
   4. Ventricular arrhythmias requiring continuous therapy, or
   5. Supraventricular arrhythmias including atrial fibrillation, which are uncontrolled.
6. Major surgery, excluding skin biopsies and procedures for insertion of central venous access devices, within 28 days prior to the start of COTI-2.
7. Active, uncontrolled bacterial, viral, fungal, or other opportunistic infection requiring systemic therapy.
8. Part 2:

   1. The presence of or imminent occurrence of airway obstruction, unless tracheostomy in place.
   2. HPV-positive status ( In HNSCC patients only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2015-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Number of dose limiting Toxicities | 12 months
  Used to measure safety and tolerability of COTI2
Tmax | 6 months
  To determine maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D)

SECONDARY OUTCOMES:
Clinical response | 6 Months
  This will be assessed through CT imaging, measurement using RECIST 1.0 criteria and GCIG criteria (if applicable)
Progression Free survival | 12 months
  This will be assessed through CT imaging and measurement using RECIST 1.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Westin, MD, Principal Investigator — MD Anderson
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrews S, von Gruenigen VE. Management of the late effects of treatments for gynecological cancer. Curr Opin Oncol. 2013 Sep;25(5):566-70. doi: 10.1097/CCO.0b013e328363e11a. PMID 23942302
- [Background] Cancer Genome Atlas Research Network. Integrated genomic analyses of ovarian carcinoma. Nature. 2011 Jun 29;474(7353):609-15. doi: 10.1038/nature10166. PMID 21720365
- [Background] Clarke MF, Dick JE, Dirks PB, Eaves CJ, Jamieson CH, Jones DL, Visvader J, Weissman IL, Wahl GM. Cancer stem cells--perspectives on current status and future directions: AACR Workshop on cancer stem cells. Cancer Res. 2006 Oct 1;66(19):9339-44. doi: 10.1158/0008-5472.CAN-06-3126. Epub 2006 Sep 21. No abstract available. PMID 16990346
- [Background] Creasman WT, Odicino F, Maisonneuve P, Quinn MA, Beller U, Benedet JL, Heintz AP, Ngan HY, Pecorelli S. Carcinoma of the corpus uteri. FIGO 26th Annual Report on the Results of Treatment in Gynecological Cancer. Int J Gynaecol Obstet. 2006 Nov;95 Suppl 1:S105-43. doi: 10.1016/S0020-7292(06)60031-3. No abstract available. PMID 17161155
- [Background] Dellinger TH, Monk BJ. Systemic therapy for recurrent endometrial cancer: a review of North American trials. Expert Rev Anticancer Ther. 2009 Jul;9(7):905-16. doi: 10.1586/era.09.54. PMID 19589030
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Freed-Pastor WA, Prives C. Mutant p53: one name, many proteins. Genes Dev. 2012 Jun 15;26(12):1268-86. doi: 10.1101/gad.190678.112. PMID 22713868
- [Background] Hirte HW, Strychowsky JE, Oliver T, Fung-Kee-Fung M, Elit L, Oza AM. Chemotherapy for recurrent, metastatic, or persistent cervical cancer: a systematic review. Int J Gynecol Cancer. 2007 Nov-Dec;17(6):1194-204. doi: 10.1111/j.1525-1438.2007.00900.x. Epub 2007 Jun 1. PMID 17540006
- [Background] Kalsi JK, Manchanda R, Menon U. Screening for gynecological cancers. Expert Rev Obstet Gynecol 2013;8(2):143-60.
- [Background] Kandoth C, McLellan MD, Vandin F, Ye K, Niu B, Lu C, Xie M, Zhang Q, McMichael JF, Wyczalkowski MA, Leiserson MDM, Miller CA, Welch JS, Walter MJ, Wendl MC, Ley TJ, Wilson RK, Raphael BJ, Ding L. Mutational landscape and significance across 12 major cancer types. Nature. 2013 Oct 17;502(7471):333-339. doi: 10.1038/nature12634. PMID 24132290
- [Background] Leary A, Auclin E, Pautier P, Lhommé C. The PI3K/Akt/mTOR pathway in ovarian cancer: biological rationale and therapeutic opportunities. In: Ovarian cancer - a clinical and translational update. InTech; 2013, pp. 275-302.
- [Background] Maleki Vareki S, Salim KY, Danter WR, Koropatnick J. Novel anti-cancer drug COTI-2 synergizes with therapeutic agents and does not induce resistance or exhibit cross-resistance in human cancer cell lines. PLoS One. 2018 Jan 24;13(1):e0191766. doi: 10.1371/journal.pone.0191766. eCollection 2018. PMID 29364966